CLINICAL TRIAL: NCT04157465
Title: Early Empirical Versus Pre-emptive Systemic Anti-fungal Therapy in Acute-on-Chronic Liver Failure Patients With Suspected Invasive Fungal Infections: a Randomized Controlled Trial
Brief Title: Anti-fungal Strategies in Acute-on-Chronic Liver Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Dr. Nipun Verma, Additional Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PGI/IEC/2019/001924
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2024-12

CONDITIONS: Antifungal Agents; Invasive Fungal Infections; Mycoses; Acute-On-Chronic Liver Failure
Keywords: cirrhosis; Acute-On-Chronic Liver Failure; liposomal amphotericin B; Invasive Fungal Infections; empiric antifungal; pre-emptive antifungal
MeSH Terms: conditions — Invasive Fungal Infections; Mycoses; Acute-On-Chronic Liver Failure; Fibrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-center, prospective randomized, open-labeled with blinded end-point (PROBE) assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Empiric group (Other): Participants will receive standard medical therapy along with the empiric strategy of treatment of invasive fungal infection (based on both risk factors and clinical suspicion of invasive fungal infection). The choice of drug will be as per institutional protocol i.e. Injection Liposomal Amphotericin B, 3-5 mg/kg of body weight as a 4- hour infusion in 5% dextrose solution. The infusion will be prepared ten minutes prior to administration by reconstituting the vial in dextrose solution by a Registered Nurse. Each vial contains 50 mg (50000U) encapsulated in liposomes. After reconstitution, the concentrate will contain 4mg/ml of the drug. During the first dose administration, 1mg will be administered with a micro drip set over ten minutes and then stopped to look for any reactions for 30 minutes. If there are no reactions, the rest of the drug is administered over 30-60 minutes period.
  Interventions: Other: Treatment strategy trial
- Pre-emptive group (Active Comparator): Participants will receive standard medical therapy along with the pre-emptive strategy of treatment of invasive fungal infection (based on risk factors, clinical suspicion and radiological or mycological evidence of invasive fungal infection). The choice of drug will be as per institutional protocol i.e. Injection Liposomal Amphotericin B, 3-5 mg/kg of body weight as a 4- hour infusion in 5% dextrose solution. The infusion will be prepared ten minutes prior to administration by reconstituting the vial in dextrose solution by a Registered Nurse. Each vial contains 50 mg (50000U) encapsulated in liposomes. After reconstitution, the concentrate will contain 4mg/ml of the drug. During the first dose administration, 1mg will be administered with a micro drip set over ten minutes and then stopped to look for any reactions for 30 minutes. If there are no reactions, the rest of the drug is administered over 30-60 minutes period.
  Interventions: Other: Treatment strategy trial

INTERVENTIONS:
Other: Treatment strategy trial — Participants will be randomly allocated in a 1:1 ratio after meeting eligibility criteria to either early empiric or pre-emptive strategy of treatment with antifungals. The antifungal treatment initiation will be at the time of allocation in the empiric group. The treatment initiation rules in the pre-emptive group will include
  1. Fungal Biomarkers positivity (Beta-D Glucan>150 pg/ml, Galactomannan index>1.0)
  2. Mycological evidence of fungal infection on fungal cultures from a non-sterile site
  3. Radiological evidence of fungal infection
  4. Other Investigations suggestive of fungal infection viz. endophthalmitis, vegetations suspicious of fungal infection, Vegetations on echocardiography with negative blood cultures for bacteria that is non-responsive to appropriate antibiotics, refractory culture-negative spontaneous bacterial peritonitis
  Treatment duration will be guided by serum biomarkers (BDG and GM) and fungal cultures.

SUMMARY:
Early treatment of invasive fungal infections (IFI) may prevent undue mortality in acute on chronic liver failure (ACLF) patients. We aim to study the impact of early empiric treatment (based on clinical suspicion) of IFI as compared to pre-emptive treatment (based on biomarkers and culture positivity) on the outcomes in ACLF patients with suspected IFI in a randomized trial. The ACLF patients with clinically suspected IFI would be randomly allocated to empiric treatment or pre-emptive treatment group and followed up clinically to assess the impact on survival, clinical outcomes and cost-effectiveness and safety of such an approach. The protocol is designed to cut- down unnecessary usage and to curtail the duration of antifungals use in ICUs based on biomarkers/culture-driven stoppage rules. The results will fuel further studies on formal cost-effective analysis and antimicrobial stewardship protocols in ACLF patients.

DETAILED DESCRIPTION:
Research question: Does an early empiric antifungal therapy improve 28-day overall survival as compared to pre-emptive antifungal therapy in critically ill, non-neutropenic adult ACLF patients with suspected IFI?

This study will be a single-center prospective randomized open-label with blinded end-point PROBE assessment and conducted at Liver ICU.

ACLF patients aged 18 to 75 years with all three criteria will be included

1. ICU stay of 48 hours or recent hospitalization
2. Two or more risk factors for IFI 3. Clinical suspicion of IFI

Exclusion criteria A Neutrophil count of less than 500 per mm3 B Recent antifungal treatment in the past 1months C Hepatocellular carcinoma or other active malignancy D Known hypersensitivity or contraindication to Liposomal AmB E HIV positivity or on HAART F Pregnancy or lactation G Moribund patients

Eligible patients will be randomly assigned, in a 1:1 ratio to receive either early empiric systemic antifungal therapy (SAT: based on risk factors and clinical suspicion) or Pre-emptive SAT (based on risk factors, clinical suspicion and radiological/investigation based evidence of fungal infection) in addition to standard medical therapy SMT and followed up for a period of 28-days or transplant or death

Empirical therapy will be Liposomal AmB 3 to 5 mg per kg of body weight per day.

It is preferred because of maximum efficacy, widest spectrum, and safety in liver disease

Pre-emptive therapy with liposomal AmB will be given if the treatment initiation rules are met including fungal biomarkers positivity, Mycological or radiological evidence of IFI

Proven-IFI will be treated as per IDSA or ESCMID guidelines in either group Stoppage rules in both groups will be based on fungal biomarkers and cultures that will be done twice weekly and twice negative bio-markers or fungal cultures at day7 and 10 will be essential to stop treatment

In case of intolerable adverse effects or contraindications to LipoAmB, the patients will undergo treatment as per IDSA guidelines Standard Medical Therapy will be as indicated and will include nutritional support, rifaximin lactulose albumin diuretics proton-pump inhibitors multivitamins and antibiotics

Outcomes will include survival at 28-day, clinical outcomes, cost-effectiveness and safety of two approaches of antifungal therapy

ELIGIBILITY:
Inclusion Criteria (All three must be present):

1. ICU stay >48 hours or admission in a tertiary care hospital prior to the current admission
2. Two or more risk factors for IFI from amongst the following:-

   1. Mechanically ventilated at least ≥ 48 hours
   2. Treatment with broad-spectrum antibacterial agents for more than 3 days
   3. Arterial or central vein catheter ≥ 2days
   4. Diabetes Mellitus
   5. Total parenteral nutrition ≥ 48 hours
   6. Acute renal failure requiring any form of renal replacement therapy ≥48hours
   7. Pancreatitis related hospitalization > 7days in last 3 months
   8. Steroid use, immunosuppressant use in the preceding 30 days
   9. High disease score as defined as MELD≥20 or APACHE II ≥16
   10. Refractory ascites, norfloxacin prophylaxis
   11. Gastrointestinal tract surgery, abdominal perforation or anastomotic leaks or any invasive procedures or surgeries in the last 7days
   12. Chronic pulmonary diseases including COPD or Tuberculosis
   13. Moderate to severe sarcopenia as defined by The Royal Free Hospital-global assessment (RFH-GA) scale60 (As per Appendix "4" )
   14. Firm diagnosis of H1N1 influenza infection in the last 3 months
3. Clinical suspicion of IFI as defined by any of the following:

   1. Evidence of unresolved sepsis/SIRS(≥ 2/4) despite appropriate broad-spectrum antibiotics beyond 3days
   2. Recrudescence of fever after a period of defervescence of at least 48 hours while still on antibiotics and without other apparent cause
   3. Tracheobronchial ulcer, nodule, plaque or pseudo-membrane
   4. Sino-nasal infection: features of acute sinusitis with at least 1 of acute localized pain, nasal ulcer, eschar, orbital involvement or
   5. Respiratory symptoms:

      * Worsening respiratory insufficiency despite appropriate ventilator support and antibiotics
      * Any 2 of Pleuritic chest pain, pleural rub, dyspnea, hemoptysis
   6. Characteristic skin lesions suspected of fungal infection
   7. Unexplained worsening of encephalopathy after initial improvement

Exclusion Criteria:

1. Neutrophil count of less than 500/mm3
2. Current or recent antifungal treatment in the past 1 months
3. Hepatocellular carcinoma or other active malignancy
4. Known hypersensitivity or contraindication to Liposomal AmB or any other AmB preparation
5. Human immunodeficiency virus seropositivity on rapid card test/ELISA, or currently on combination antiretroviral therapy (cART)
6. Pregnancy as confirmed by urine pregnancy test or lactation
7. Moribund patients as defined as

   1. ≥ 4 organ failure as per CLIF-SOFA score
   2. Signs of brainstem death- absent brainstem reflexes
   3. Expected ICU stay <48 hours

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 28 day
  28-day overall survival

SECONDARY OUTCOMES:
Incidence of proven or probable IFI | 28 day
  Incidence of proven or probable IFI at 28 days
In-hospital mortality | 28 day
  Number of participants dying in hospital due to any cause within 28 day of enrollment
Evolution of organ failures as assessed by chronic liver failure-sequential organ failure score (CLIF-SOFA) | 28 day
  Development of new or worsening organ failures as defined by chronic liver failure -sequential organ failure (CLIF-SOFA) scores within 28 days of enrollment. CLIF-SOFA score ranges from 0-24 incorporating 6 organ systems and 0 being best and 24 being worst.
Evolution of serum 1, 3 Beta-D Glucan (BDG; in pg/ml) levels throughout the study period | 28 day
  Trends of 1, 3 Beta-D Glucan (BDG) throughout the study period that will be done on twice weekly intervals after enrollment
Evolution of serum Galactomannan index (GM; in %) throughout the study period | 28 day
  Trends of Galactomannan index (GM; in %) throughout the study period that will be done on twice weekly intervals after enrollment
Incidence of key events like new onset ventilator associated pneumonia, urinary tract infection, spontaneous fungal peritonitis | 28 day
  Incidence of key events like new onset VAP, UTI, fungal SBP
Mechanical ventilation free days | 28 day
  Duration free from mechanical ventilation within 28 days of enrollment
Length of ICU and hospital stay | 28 day
  Effect on length of ICU, hospital stay within 28 day of enrollment
Treatment success rate | 28 day
  Treatment success rate, successful treatment being defined as
  1. Survival beyond 7 days of start of SAT with resolution of sepsis attributable to IFI
  2. Absence of new/ breakthrough IFI during treatment or within 7 days of completion
  3. Absence of treatment discontinuation related to toxicity/lack of efficacy

OTHER OUTCOMES:
Number of participants with adverse events due to antifungals requiring cessation of therapy | 28 day
  Number of participants out of whole group who would develop adverse events due to antifungals that will require cessation of therapy within 28 day of enrollment
Out of pocket expenditure | 28 day
  Out of pocket expenditure incurred by the patients in two groups

CONTACTS AND LOCATIONS:
Overall Officials: Nipun Verma, MD, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical education and Research, Chandigarh, Uttarakhand, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verma N, Valsan A, Garg P, Sarabu S, Kaur P, Mohan N, De A, Premkumar M, Taneja S, Prinja S, Chakrabarti A, Shafiq N, Duseja A. Empirical Antifungal Therapy Improves Survival in Patients With Acute-on-Chronic Liver Failure With Suspected Invasive Fungal Infections: A Pragmatic Randomized Trial. Am J Gastroenterol. 2025 Nov 21. doi: 10.14309/ajg.0000000000003832. Online ahead of print. PMID 41268913